CLINICAL TRIAL: NCT05726708
Title: Impact of an E-Learning Parental Coaching for Parents of Young Children With Autism Spectrum Disorder
Brief Title: Impact of an E-Learning Coaching for Parents of Young Children With Autism
Acronym: ECOACH
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Vaudois (Other)
Responsible Party: Principal Investigator, Nadia Chabane, Professor, Centre Hospitalier Universitaire Vaudois
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 552
Record Dates: First submitted 2023-01-26; First posted 2023-02-14 (Actual); Last update posted 2024-02-08 (Actual); Status verified 2024-02

CONDITIONS: Autism Spectrum Disorder
Keywords: autism; parental coaching
MeSH Terms: conditions — Autism Spectrum Disorder; Autistic Disorder

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- E-Learning (Experimental): E-Learning coaching. 11 modules on line. 5 debriefing on visio conference with a professional (1/month)
  Interventions: Behavioral: E-Learning
- Paediatric Autism Communication Therapy (PACT) (Active Comparator): Parents will have 12 coaching sessions with a therapist, following the PACT model. Between each session, the parent will be asked to practice the strategies at home and to film themselves doing an activity with their child (10-minute film).
  Interventions: Behavioral: E-Learning
- Control (No Intervention): No parental coaching

INTERVENTIONS:
Behavioral: E-Learning — On line modules of coaching for parents
  Arms: E-Learning; Paediatric Autism Communication Therapy (PACT)

SUMMARY:
The goal of this study is to evaluate the impact of a parental coaching based on E-Learning (EL), intended for parents of children with autism spectrum disorder (ASD). Population: parents of young children (2 to 4 years old) with an ASD diagnosis.

The main questions that our study will answer are:

* Has parental coaching via E-Learning a significant impact compared to no coaching?
* If so, is that impact comparable to standard parental coaching such as PACT?

The impact will be evaluated in three domains:

* Child development: behavior, sleep, eating behavior
* Parental competences: stress, coping, feeling of parental competencies
* Parent-child interaction: communication, visual attention

The investigators will compare 3 groups:

1. ASD children whose parents will follow a parental coaching via E-learning,
2. ASD children whose parents will follow a standard parental coaching (PACT)
3. ASD children whose parents will not follow any specific coaching program

ELIGIBILITY:
Inclusion Criteria:

* Children with ASD
* Age 2 years to 4 years and 6 months
* Family speaking french
* Parent who signed the consent form

Exclusion Criteria:

* children with known genetic syndrome
* children with visual or auditive deficit
* children with epilepsy
* no internet access
* no french speaking

Ages: 24 Months to 48 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 99 (Estimated)
Dates: Start 2023-10-24 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Dyadic Communication Measure for Autism (DCMA) before parental coaching | Month 0
  DCMA is a measure of the natural flowing dyadic communication interaction between parent and child in a free play context. It was originally designed to capture aspects of communication in young children with autism and aspects of the parent communication style that are often targeted in communication-focussed interventions. It Is grounded in the theory and research on pragmatic language development in children, specifically in children with autism. DCMA involves video-recording the parent and child playing together in a natural way using a standard set of toys. The interaction is then coded from video-tape and three levels of the interaction are observed:
  * Parent synchrony and responsiveness
  * Child communicative initiations, responses and communicative functions
  * Amount of mutual shared attention between parent and child
Dyadic Communication Measure for Autism (DCMA) immediately after the end of parental coaching | Month 6
  DCMA is a measure of the natural flowing dyadic communication interaction between parent and child in a free play context. It was originally designed to capture aspects of communication in young children with autism and aspects of the parent communication style that are often targeted in communication-focussed interventions. It Is grounded in the theory and research on pragmatic language development in children, specifically in children with autism. DCMA involves video-recording the parent and child playing together in a natural way using a standard set of toys. The interaction is then coded from video-tape and three levels of the interaction are observed:
  * Parent synchrony and responsiveness
  * Child communicative initiations, responses and communicative functions
  * Amount of mutual shared attention between parent and child
Dyadic Communication Measure for Autism (DCMA) 6 months after the end of parental coaching | Month 12
  DCMA is a measure of the natural flowing dyadic communication interaction between parent and child in a free play context. It was originally designed to capture aspects of communication in young children with autism and aspects of the parent communication style that are often targeted in communication-focussed interventions. It Is grounded in the theory and research on pragmatic language development in children, specifically in children with autism. DCMA involves video-recording the parent and child playing together in a natural way using a standard set of toys. The interaction is then coded from video-tape and three levels of the interaction are observed:
  * Parent synchrony and responsiveness
  * Child communicative initiations, responses and communicative functions
  * Amount of mutual shared attention between parent and child
Brief Observation of Social Communication Change (BOSCC) before parental coaching | Month 0
  BOSCC is a treatment response measure of autism spectrum disorder (ASD) symptoms. The BOSCC is a behavioral coding scheme that is applied to 10-12 min videotaped social/play interactions between a child and a researcher or caregiver (play partner). The coding scheme was developed by expanding items from the Autism Diagnostic Observation Schedule (ADOS), to quantify more nuanced variation in ASD symptoms.
Brief Observation of Social Communication Change (BOSCC) immediately after the end of parental coaching | Month 6
  BOSCC is a treatment response measure of autism spectrum disorder (ASD) symptoms. The BOSCC is a behavioral coding scheme that is applied to 10-12 min videotaped social/play interactions between a child and a researcher or caregiver (play partner). The coding scheme was developed by expanding items from the Autism Diagnostic Observation Schedule (ADOS), to quantify more nuanced variation in ASD symptoms.
Brief Observation of Social Communication Change (BOSCC) 6 months after the end of parental coaching | Month 12
  BOSCC is a treatment response measure of autism spectrum disorder (ASD) symptoms. The BOSCC is a behavioral coding scheme that is applied to 10-12 min videotaped social/play interactions between a child and a researcher or caregiver (play partner). The coding scheme was developed by expanding items from the Autism Diagnostic Observation Schedule (ADOS), to quantify more nuanced variation in ASD symptoms.
Percentage of synchronized communication acts with the parents and professionals before parental coaching | Month 0
  Head-mounted Eye tracking system to record eye movements during Dyadic Communication Measure for Autism (DCMA) and Brief Observation of Social Communication Change (BOSCC). Head-mounted eye trackers not only capture the child's view of their environment, but also track where they are looking in first person, at all times, allowing us to study gaze in more naturalistic situations. In particular, wearable eye trackers improve the construct validity of developmentally important concepts, such as visual object experiences and social attention, in ways that would be impossible with screen-based eye trackers. The investigators will measure the percentage of synchronous communication acts with the parents and professionals.
Percentage of synchronized communication acts with the parents and professionals immediately after the end of parental coaching | Month 6
  Head-mounted Eye tracking system to record eye movements during Dyadic Communication Measure for Autism (DCMA) and Brief Observation of Social Communication Change (BOSCC). Head-mounted eye trackers not only capture the child's view of their environment, but also track where they are looking in first person, at all times, allowing us to study gaze in more naturalistic situations. In particular, wearable eye trackers improve the construct validity of developmentally important concepts, such as visual object experiences and social attention, in ways that would be impossible with screen-based eye trackers. The investigators will measure the percentage of synchronous communication acts with the parents and professionals.
Percentage of synchronized communication acts with the parents and professionals 6 months after the end of parental coaching | Month 12
  Head-mounted Eye tracking system to record eye movements during Dyadic Communication Measure for Autism (DCMA) and Brief Observation of Social Communication Change (BOSCC). Head-mounted eye trackers not only capture the child's view of their environment, but also track where they are looking in first person, at all times, allowing us to study gaze in more naturalistic situations. In particular, wearable eye trackers improve the construct validity of developmentally important concepts, such as visual object experiences and social attention, in ways that would be impossible with screen-based eye trackers. The investigators will measure the percentage of synchronous communication acts with the parents and professionals.
Mullen Scales of Early Learning (MSEL) before parental coaching | Month 0
  The Mullen Scales of Early Learning (MSEL) is a standardized assessment commonly used in clinical psychology as a developmental measure of cognitive development in children 2 to 5½ years of age. The MSEL is organized into 5 subscales: (a) gross motor, (b) fine motor, (c) visual reception (or non-verbal problem solving), (d) receptive language, and (e) expressive language. An early learning composite score can be derived from fine motor, visual reception, receptive language, and expressive language scales. For young children this early learning composite score is considered equivalent to a more traditional intelligence quotient score or a developmental standard score. Each subscale is standardized to calculate a standard score, percentile and age-equivalent score. The maximum achievable raw score per scale is 50 for the visual reception scale, 49 for the fine motor scale, 48 for the receptive language scale and 50 for the expressive language scale. Higher scores mean a better outcome.
Mullen Scales of Early Learning (MSEL) immediately after the end of parental coaching | Month 6
  The Mullen Scales of Early Learning (MSEL) is a standardized assessment commonly used in clinical psychology as a developmental measure of cognitive development in children 2 to 5½ years of age. The MSEL is organized into 5 subscales: (a) gross motor, (b) fine motor, (c) visual reception (or non-verbal problem solving), (d) receptive language, and (e) expressive language. An early learning composite score can be derived from fine motor, visual reception, receptive language, and expressive language scales. For young children this early learning composite score is considered equivalent to a more traditional intelligence quotient score or a developmental standard score. Each subscale is standardized to calculate a standard score, percentile and age-equivalent score. The maximum achievable raw score per scale is 50 for the visual reception scale, 49 for the fine motor scale, 48 for the receptive language scale and 50 for the expressive language scale. Higher scores mean a better outcome.
Mullen Scales of Early Learning (MSEL) 6 months after the end of parental coaching | Month 12
  The Mullen Scales of Early Learning (MSEL) is a standardized assessment commonly used in clinical psychology as a developmental measure of cognitive development in children 2 to 5½ years of age. The MSEL is organized into 5 subscales: (a) gross motor, (b) fine motor, (c) visual reception (or non-verbal problem solving), (d) receptive language, and (e) expressive language. An early learning composite score can be derived from fine motor, visual reception, receptive language, and expressive language scales. For young children this early learning composite score is considered equivalent to a more traditional intelligence quotient score or a developmental standard score. Each subscale is standardized to calculate a standard score, percentile and age-equivalent score. The maximum achievable raw score per scale is 50 for the visual reception scale, 49 for the fine motor scale, 48 for the receptive language scale and 50 for the expressive language scale. Higher scores mean a better outcome.
Child Eating Behaviour Questionnaire (CEBQ) before parental coaching | Month 0
  CEBQ is a 35-item parent-report questionnaire assessing eating style in children. Eating style is assessed on eight scales: food responsiveness (4 items), enjoyment of food (4 items), emotional overeating (4 items), desire to drink (3 items), satiety responsiveness (5 items), slowness in eating (4 items), and emotional undereating (4 items), and fussiness (7 items). Informants rate the frequency of their child's behaviors and experiences on a 5-point scale: 1 = never, 2 = rarely, 3 = sometimes, 4 = often, 5 = always.
Child Eating Behaviour Questionnaire (CEBQ) immediately after the end of parental coaching | Month 6
  CEBQ is a 35-item parent-report questionnaire assessing eating style in children. Eating style is assessed on eight scales: food responsiveness (4 items), enjoyment of food (4 items), emotional overeating (4 items), desire to drink (3 items), satiety responsiveness (5 items), slowness in eating (4 items), and emotional undereating (4 items), and fussiness (7 items). Informants rate the frequency of their child's behaviors and experiences on a 5-point scale: 1 = never, 2 = rarely, 3 = sometimes, 4 = often, 5 = always.
Child Eating Behaviour Questionnaire (CEBQ) 6 months after the end of parental coaching | Month 12
  CEBQ is a 35-item parent-report questionnaire assessing eating style in children. Eating style is assessed on eight scales: food responsiveness (4 items), enjoyment of food (4 items), emotional overeating (4 items), desire to drink (3 items), satiety responsiveness (5 items), slowness in eating (4 items), and emotional undereating (4 items), and fussiness (7 items). Informants rate the frequency of their child's behaviors and experiences on a 5-point scale: 1 = never, 2 = rarely, 3 = sometimes, 4 = often, 5 = always.
Child Behavior Checklist (CBCL)/1.5-5 before parental coaching | Month 0
  The CBCL/1.5-5 obtains caregivers' ratings of 99 problem items. Items are scored on the following syndrome scales: Emotionally Reactive, Anxious/Depressed, Somatic Complaints, Withdrawn, Attention Problems, Aggressive Behavior, and Sleep Problems. Items are also scored on the following Diagnostic and Statistical Manual (DSM)-oriented scales: Affective Problems, Anxiety Problems, Pervasive Developmental Problems, Attention Deficit/Hyperactivity Problems, Stress Problems, Autism Spectrum Problems, and Oppositional Defiant Problems. According to the normative data of the CBCL, a t-score ≤ 59 indicates non-clinical symptoms, a t-score between 60 and 64 indicates that the child is at risk for problem behaviors, and a t-score ≥ 65 indicates clinical symptoms. Higher scores mean thus a worse outcome.
Child Behavior Checklist (CBCL)/1.5-5 immediately after the end of parental coaching | Month 6
  The CBCL/1.5-5 obtains caregivers' ratings of 99 problem items. Items are scored on the following syndrome scales: Emotionally Reactive, Anxious/Depressed, Somatic Complaints, Withdrawn, Attention Problems, Aggressive Behavior, and Sleep Problems. Items are also scored on the following Diagnostic and Statistical Manual (DSM)-oriented scales: Affective Problems, Anxiety Problems, Pervasive Developmental Problems, Attention Deficit/Hyperactivity Problems, Stress Problems, Autism Spectrum Problems, and Oppositional Defiant Problems. According to the normative data of the CBCL, a t-score ≤ 59 indicates non-clinical symptoms, a t-score between 60 and 64 indicates that the child is at risk for problem behaviors, and a t-score ≥ 65 indicates clinical symptoms. Higher scores mean thus a worse outcome.
Child Behavior Checklist (CBCL)/1.5-5 6 months after the end of parental coaching | Month 12
  The CBCL/1.5-5 obtains caregivers' ratings of 99 problem items. Items are scored on the following syndrome scales: Emotionally Reactive, Anxious/Depressed, Somatic Complaints, Withdrawn, Attention Problems, Aggressive Behavior, and Sleep Problems. Items are also scored on the following Diagnostic and Statistical Manual (DSM)-oriented scales: Affective Problems, Anxiety Problems, Pervasive Developmental Problems, Attention Deficit/Hyperactivity Problems, Stress Problems, Autism Spectrum Problems, and Oppositional Defiant Problems. According to the normative data of the CBCL, a t-score ≤ 59 indicates non-clinical symptoms, a t-score between 60 and 64 indicates that the child is at risk for problem behaviors, and a t-score ≥ 65 indicates clinical symptoms. Higher scores mean thus a worse outcome.
Paediatric Sleep questionnaire (PSQ) before parental coaching | Month 0
  PSQ contains 22 symptom items that ask about snoring frequency, loud snoring, observed apneas, difficulty breathing during sleep, daytime sleepiness, inattentive or hyperactive behavior, and other pediatric sleep-related features. Subscales within the PSQ include a 4-item sleepiness scale, a 4-item snoring scale, and a 6-item in attention/hyperactivity scale. The answers are scored as "0" (symptom absent) or "1" (symptom present) and the overall score is calculated as a proportion of positive answers with a score greater or equal to 0.33 being considered predictive for sleep disordered breathing. Higher scores mean thus a worse outcome.
Paediatric Sleep questionnaire (PSQ) immediately after the end of parental coaching | Month 6
  PSQ contains 22 symptom items that ask about snoring frequency, loud snoring, observed apneas, difficulty breathing during sleep, daytime sleepiness, inattentive or hyperactive behavior, and other pediatric sleep-related features. Subscales within the PSQ include a 4-item sleepiness scale, a 4-item snoring scale, and a 6-item in attention/hyperactivity scale. The answers are scored as "0" (symptom absent) or "1" (symptom present) and the overall score is calculated as a proportion of positive answers with a score greater or equal to 0.33 being considered predictive for sleep disordered breathing. Higher scores mean thus a worse outcome.
Paediatric Sleep questionnaire (PSQ) 6 months after the end of parental coaching | Month 12
  PSQ contains 22 symptom items that ask about snoring frequency, loud snoring, observed apneas, difficulty breathing during sleep, daytime sleepiness, inattentive or hyperactive behavior, and other pediatric sleep-related features. Subscales within the PSQ include a 4-item sleepiness scale, a 4-item snoring scale, and a 6-item in attention/hyperactivity scale. The answers are scored as "0" (symptom absent) or "1" (symptom present) and the overall score is calculated as a proportion of positive answers with a score greater or equal to 0.33 being considered predictive for sleep disordered breathing. Higher scores mean thus a worse outcome.
Parenting Stress Index (PSI) before parental coaching | Month 0
  PSI is a questionnaire designed to measure the extent of stress in the parent-child relationship. This diagnostic instrument is based on the assumption that the integral stress experienced by the parent depends on certain characteristics of the child, the parent, and the parenting situation. Child stress features are measured on six scales:
  Hyperactivity/Distraction, Adaptability, Reinforcement, Demands, Mood, Acceptability. Parent personality and situational variables are measured on seven scales: Depression, Sense of competence, Attachment, Marital relationship, Social isolation, Parenting health, Parenting restrictions. PSI has 36 items based on a five-point Likert scale where each value corresponds to a specific statement (1 = completely disagree; 5 = completely agree). The subscale scores range from 12 to 60, and the Total Stress score ranges from 36 to 180. The higher the score, the greater the level of parental stress.
Parenting Stress Index (PSI) immediately after the end of parental coaching | Month 6
  PSI is a questionnaire designed to measure the extent of stress in the parent-child relationship. This diagnostic instrument is based on the assumption that the integral stress experienced by the parent depends on certain characteristics of the child, the parent, and the parenting situation. Child stress features are measured on six scales:
  Hyperactivity/Distraction, Adaptability, Reinforcement, Demands, Mood, Acceptability. Parent personality and situational variables are measured on seven scales: Depression, Sense of competence, Attachment, Marital relationship, Social isolation, Parenting health, Parenting restrictions. PSI has 36 items based on a five-point Likert scale where each value corresponds to a specific statement (1 = completely disagree; 5 = completely agree). The subscale scores range from 12 to 60, and the Total Stress score ranges from 36 to 180. The higher the score, the greater the level of parental stress.
Parenting Stress Index (PSI) 6 months after the end of parental coaching | Month 12
  PSI is a questionnaire designed to measure the extent of stress in the parent-child relationship. This diagnostic instrument is based on the assumption that the integral stress experienced by the parent depends on certain characteristics of the child, the parent, and the parenting situation. Child stress features are measured on six scales:
  Hyperactivity/Distraction, Adaptability, Reinforcement, Demands, Mood, Acceptability. Parent personality and situational variables are measured on seven scales: Depression, Sense of competence, Attachment, Marital relationship, Social isolation, Parenting health, Parenting restrictions. PSI has 36 items based on a five-point Likert scale where each value corresponds to a specific statement (1 = completely disagree; 5 = completely agree). The subscale scores range from 12 to 60, and the Total Stress score ranges from 36 to 180. The higher the score, the greater the level of parental stress.
Parenting Sense of Competence Scale (PSOC) before parental coaching | Month 0
  The PSOC questionnaire is composed of 17 statements that measure the feeling of competence in the exercise of the parental role. It has two subscales: seven statements concern the feeling of efficacy and ten others, the feeling of satisfaction. One version is available for the father and another for the mother. Respondents rate their parenting competence on a six-point Likert-type scale ranging from "strongly agree" (1) to "strongly disagree" (6). The score can vary from 7 to 42, with a score of 7 to 13 indicating a very low sense of efficacy and a score of 38 to 42 indicating a very high sense of efficacy on the continuum. Higher scores mean thus a better outcome.
Parenting Sense of Competence Scale (PSOC) immediately after the end of parental coaching | Month 6
  The PSOC questionnaire is composed of 17 statements that measure the feeling of competence in the exercise of the parental role. It has two subscales: seven statements concern the feeling of efficacy and ten others, the feeling of satisfaction. One version is available for the father and another for the mother. Respondents rate their parenting competence on a six-point Likert-type scale ranging from "strongly agree" (1) to "strongly disagree" (6). The score can vary from 7 to 42, with a score of 7 to 13 indicating a very low sense of efficacy and a score of 38 to 42 indicating a very high sense of efficacy on the continuum. Higher scores mean thus a better outcome.
Parenting Sense of Competence Scale (PSOC) 6 months after the end of parental coaching | Month 12
  The PSOC questionnaire is composed of 17 statements that measure the feeling of competence in the exercise of the parental role. It has two subscales: seven statements concern the feeling of efficacy and ten others, the feeling of satisfaction. One version is available for the father and another for the mother. Respondents rate their parenting competence on a six-point Likert-type scale ranging from "strongly agree" (1) to "strongly disagree" (6). The score can vary from 7 to 42, with a score of 7 to 13 indicating a very low sense of efficacy and a score of 38 to 42 indicating a very high sense of efficacy on the continuum. Higher scores mean thus a better outcome.
Child Adjustment and Parent Efficacy Scale (CAPES) before parental coaching | Month 0
  Child Adjustment and Parent Efficacy Scale (CAPES) is a parent-report questionnaire that measures child behavioural and emotional adjustment and parental efficacy. It consists of 30 items rated on a 4-point scale, ranging from not true of my child at all (0) to true of my child very much, or most of the time (3), where 20 items are two-part questions that assess both child behaviour and parent efficacy. Twenty-six items assess behaviour concerns (e.g., My child rudely answers back to me) and behavioural competencies (Behaviour Scale; e.g., My child follows rules and limits), and four items assess emotional adjustment (Emotional Maladjustment Scale; e.g., My child worries). Some items are reverse scored. Items are summed to yield a total intensity score (CAPES intensity scale: range of 0-90), which is made up of a behaviour score (range of 0-78) and an emotional maladjustment score (0-12) where high scores indicate higher levels of problems.
Child Adjustment and Parent Efficacy Scale (CAPES) immediately after the end of parental coaching | Month 6
  Child Adjustment and Parent Efficacy Scale (CAPES) is a parent-report questionnaire that measures child behavioural and emotional adjustment and parental efficacy. It consists of 30 items rated on a 4-point scale, ranging from not true of my child at all (0) to true of my child very much, or most of the time (3), where 20 items are two-part questions that assess both child behaviour and parent efficacy. Twenty-six items assess behaviour concerns (e.g., My child rudely answers back to me) and behavioural competencies (Behaviour Scale; e.g., My child follows rules and limits), and four items assess emotional adjustment (Emotional Maladjustment Scale; e.g., My child worries). Some items are reverse scored. Items are summed to yield a total intensity score (CAPES intensity scale: range of 0-90), which is made up of a behaviour score (range of 0-78) and an emotional maladjustment score (0-12) where high scores indicate higher levels of problems.
Child Adjustment and Parent Efficacy Scale (CAPES) 6 months after the end of parental coaching | Month 12
  Child Adjustment and Parent Efficacy Scale (CAPES) is a parent-report questionnaire that measures child behavioural and emotional adjustment and parental efficacy. It consists of 30 items rated on a 4-point scale, ranging from not true of my child at all (0) to true of my child very much, or most of the time (3), where 20 items are two-part questions that assess both child behaviour and parent efficacy. Twenty-six items assess behaviour concerns (e.g., My child rudely answers back to me) and behavioural competencies (Behaviour Scale; e.g., My child follows rules and limits), and four items assess emotional adjustment (Emotional Maladjustment Scale; e.g., My child worries). Some items are reverse scored. Items are summed to yield a total intensity score (CAPES intensity scale: range of 0-90), which is made up of a behaviour score (range of 0-78) and an emotional maladjustment score (0-12) where high scores indicate higher levels of problems.
Brief Coping Orientation to Problems Experienced (Brief-COPE) Inventory before parental coaching | Month 0
  The Brief Coping Orientation to Problems Experienced (Brief-COPE) is a 28 item self-report questionnaire designed to measure effective and ineffective ways to cope with a stressful life event. "Coping" is defined broadly as an effort used to minimise distress associated with negative life experiences. The scale is often used in health-care settings to ascertain how patients are emotionally responding to a serious circumstance.
  It is comprised of 14 scales, each of which assesses the degree to which a respondent utilizes a specific coping strategy. Respondents rate items on a 4-point Likert scale, ranging from 1 - "I haven't been doing this at all" to 4 - "I've been doing this a lot." Each of the 14 scales is comprised of 2 items; total scores on each scale range from 2 (minimum) to 8 (maximum). Higher scores indicate increased utilization of that specific coping strategy.
Brief Coping Orientation to Problems Experienced (Brief-COPE) Inventory immediately after the end of parental coaching | Month 6
  The Brief Coping Orientation to Problems Experienced (Brief-COPE) is a 28 item self-report questionnaire designed to measure effective and ineffective ways to cope with a stressful life event. "Coping" is defined broadly as an effort used to minimise distress associated with negative life experiences. The scale is often used in health-care settings to ascertain how patients are emotionally responding to a serious circumstance.
  It is comprised of 14 scales, each of which assesses the degree to which a respondent utilizes a specific coping strategy. Respondents rate items on a 4-point Likert scale, ranging from 1 - "I haven't been doing this at all" to 4 - "I've been doing this a lot." Each of the 14 scales is comprised of 2 items; total scores on each scale range from 2 (minimum) to 8 (maximum). Higher scores indicate increased utilization of that specific coping strategy.
Brief Coping Orientation to Problems Experienced (Brief-COPE) Inventory 6 months after the end of parental coaching | Month 12
  The Brief Coping Orientation to Problems Experienced (Brief-COPE) is a 28 item self-report questionnaire designed to measure effective and ineffective ways to cope with a stressful life event. "Coping" is defined broadly as an effort used to minimise distress associated with negative life experiences. The scale is often used in health-care settings to ascertain how patients are emotionally responding to a serious circumstance.
  It is comprised of 14 scales, each of which assesses the degree to which a respondent utilizes a specific coping strategy. Respondents rate items on a 4-point Likert scale, ranging from 1 - "I haven't been doing this at all" to 4 - "I've been doing this a lot." Each of the 14 scales is comprised of 2 items; total scores on each scale range from 2 (minimum) to 8 (maximum). Higher scores indicate increased utilization of that specific coping strategy.

CONTACTS AND LOCATIONS:
Locations (1):
- Service des troubles du spectre de l'autisme et apparentés, Lausanne, Switzerland

IPD SHARING:
Plan to Share IPD: No